CLINICAL TRIAL: NCT04084431
Title: Supportive Care With or Without Repeated Whole Brain Radiotherapy in Patients With Recurrent Brain Metastases Unsuitable for Resection or Stereotactic Radiotherapy.
Brief Title: Supportive Care With or Without Repeated Whole Brain Radiotherapy in Patients With Recurrent Brain Metastases
Acronym: RECARE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: organizational reasons
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECARE Trial Version 1.1
Record Dates: First submitted 2019-08-27; First posted 2019-09-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Brain Metastases
Keywords: repeated whole brain radiation therapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: Prospective, randomized 2-armed Phase II Pilot-Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WBRT (10 x 2 Gy) + OSC (Active Comparator): Whole brain radiotherapy will be applied with a total dose of 20 Gy in 10 fractions (single dose of 2 Gy). OSC as needed.
  Interventions: Radiation: Radiation
- Optimal Supportive Care (OSC) alone (Experimental): Symptomatic treatment including steroids, pain medication, nutritional support, etc
  Interventions: Other: OSC

INTERVENTIONS:
Radiation: Radiation — WBRT will be applied in 10 fractions with single doses of 2 Gy (Arm 1) to the whole brain
  Arms: WBRT (10 x 2 Gy) + OSC
Other: OSC — optimal supportive Care (OSC) alone
  Arms: Optimal Supportive Care (OSC) alone

SUMMARY:
Patients with solid cancers may develop cerebral metastases, requiring whole brain radiotherapy (WBRT). Furthermore, in several cases, a secondary course of WBRT might be required due to intracerebral recurrence and limited options for alternative treatments, besides optimal supportive care (OSC). There have been few reports on re-irradiation of the whole brain, but further evaluation especially of the optimal dose concept is warranted. Especially, the efficacy compared to OSC has to date not been evaluated.

The present trial aims at evaluating the efficacy of a repeated WBRT with a total dose of 20 Gy in 10 fractions compared to OSC.

Primary endpoint is time to WHO performance status (PS) deterioration to more than 3 (duration of functional independence).

Secondary endpoints are quality of life, overall survival, radiation-induced toxicity and functional independence assessed by the Barthel Index of Activities of Daily Living (ADL)1.

DETAILED DESCRIPTION:
According to Nussbaum et al., 24-45% of cancer patients develop cerebral metastases during their disease. Brain metastases are generally associated with a poor prognosis and high morbidity2. Published median survival rates after WBRT are between 2 and 7 months3. Standard of care in multiple BM is WBRT delivered as total dose of 30 Gy in 10 fractions, leading to modest palliation with a median survival of 3 to 5 months 4-6. Prognostic factors include the RPA-classification, performance status, response to steroids and evidence of systemic disease3,6.

Unfortunately, intracerebral recurrence happens 7-9. For example, in the cohort of Meyners et al. (2010) on WBRT in relatively radio-resistant tumours, median time to recurrence was 4.5 months and the local control rates at 6 and 12 months after radiotherapy were 37% and 15%, respectively10. Furthermore, the treatment of intracerebral recurrence after previous WBRT is challenging. In case of ≤ 3 recurrent BM, surgery or stereotactic radiosurgery (SRS) are options. One other option, especially in case of >3 recurrent BM is repeated WBRT. In this setting, one of the first reports on repeated WBRT was published by Cooper et al. in 199011. The authors reported on repeated WBRT (n=52) consisting of a total dose of 25 Gy in 10 fractions. Response to re-irradiation was seen in about 40% of the patients. Furthermore, the patients improved by at least one level in their neurologic function status. Survival after second therapy averaged 5 months. In the report by Wong et al. (1996) median dose of retreatment (n=86) was 20 Gy12. Resolution of symptoms was achieved in 27% of patients, partial improvement in 43% and no improvement or worsening of symptoms was seen in 29% of patients. The majority of patients had no significant toxicity in consequence of re-irradiation. Five patients had radiographic abnormalities of their brain consistent with radiation-related changes. One patient had symptoms of dementia that was thought to be caused by radiotherapy. Sadikov et al. (2007) reported on 72 patients who underwent repeated WBRT for recurrent or progressive BM13. The median survival after re-irradiation was 4.1 months. One patient was reported having memory impairment and pituitary insufficiency after 5 months of progression-free survival.

In the report by Mayer et al. on re-irradiation tolerance of the human brain (this analysis was focused on recurrent glioma), the authors concluded that radiation-induced brain tissue necrosis is likely to occur at normalized tolerance doses of cumulative > 100 Gy14.

The recent QUARTZ trial investigated the efficacy of WBRT vs. OSC in patients with non-small cell lung cancer and low performance status. The results suggest that WBRT, even in the primary situation, offers no substantial benefit to most patients with brain metastases from NSCLC in terms of improved survival, overall quality of life, or reduction of steroid use in this cohort15.

In the present trial, the primary endpoint (time to WHO PS deterioration to more than 3) as well as the secondary endpoints QoL, overall survival, radiation-induced toxicity and functional independence assessed by the Barthel Index of Activities of Daily Living (ADL) in patients previously treated with WBRT requiring repeated WBRT for intracerebral tumour progression will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed malignancy
* previous WBRT or prophylactic whole brain irradiation (PCI)
* MR- or CT-imaging confirmed recurrent cerebral metastases (>10)
* Or: MR- or CT-imaging confirmed recurrent cerebral metastases (1-10) and inability to perform SRS or surgery (e.g. meningeal carcinomatosis), concluded by interdisciplinary conference
* age ≥ 18 years
* Time between initial WBRT/PCI and recurrent WBRT >3 months
* WHO performance score ≤3
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* • refusal to take part in the study

  * Pregnant or lactating women
  * Participation in another competing clinical study or observation period of competing trials, respectively
  * Ability to perform SRS or surgery on brain metastases as a treatment alternative
  * Systemic anticancer treatment <4 weeks for chemotherapy and <1 week for TKIs and targeted therapies before randomisation.
  * Persons who are in a relationship of dependence/employment with the investigators
  * Cerebral lymphomas, metastases of germ cell tumours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to WHO PS to more than 3 | up to 4 years or from date of randomization unitl the date of documented date of death from any cause
  WHO Performance status

SECONDARY OUTCOMES:
OS | up to 4 years or from date of randomization unitl the date of documented date of death from any cause
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No